CLINICAL TRIAL: NCT05931562
Title: An Interventional Study on the Association Between Diet, Cognitive Function, Stress and the Gut Microbiota in Healthy Volunteers.
Brief Title: The Impact of Diet on the Gut-Microbiota-Brain Axis
Acronym: NMB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: APC 150b
Record Dates: First submitted 2023-06-12; First posted 2023-07-05 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Microbiota-gut-brain axis; Diet; Cognition; Stress; Dietary Fibre; Fermented foods
MeSH Terms: interventions — Fermented Foods

STUDY DESIGN:
Intervention Model Description: Randomized-controlled, parallel, single-blinded design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator): Participants will recieve dietary education based on the healthy eating guidleines provided by the Health Service Executive (HSE).
  Interventions: Other: Control
- Fermented Foods (Experimental): Fermented foods diet (4-6 portions/day)
  Interventions: Other: Fermented Foods
- High Fibre (Experimental): High fibre diet (24-35 grams/day)
  Interventions: Other: High Fibre
- Combined Diet (Experimental): Combined diet high in fibre and fermented foods (fibre aim 24-35 grams/day, fermented foods aim 4-6 portions/day)
  Interventions: Other: Combined Diet

INTERVENTIONS:
Other: Fermented Foods — Participants will recieve dietary education to include 4 to 6 portions of fermented foods to their normal diet.
  Arms: Fermented Foods
Other: High Fibre — Participants will recieve dietary education to increase their fibre intake to 24-35g/day in their normal diet.
  Arms: High Fibre
Other: Combined Diet — Participants will recieve dietary education to increase their fibre intake to 25-30g/day and include 3 to 4 portions of fermented foods to their normal diet.
  Arms: Combined Diet
Other: Control — Participants will recieve dietary education based on the Irish healthy food pyramid.
  Arms: Control

SUMMARY:
This study aims to investigate the effects of an 8-week dietary intervention on cognitive function, stress, and the gut microbiota in healthy adults with low fibre intake.

DETAILED DESCRIPTION:
The gut microbiota communicates bidirectionally with the brain via the microbiota-gut-brain axis to influence various aspects of human physiology, including host metabolism, immune function, behaviour, and cognition. Diet is a key modulator of the microbial composition, suggesting that the microbiota could explain the association between poor nutrition and decreasing health of the population. Dietary fibre is the main energy source for the gut microbiota and fundamentally impacts its composition and function. The microbiota-gut-brain axis has been proposed to mediate some of the effects of dietary fibre on the brain, for example through microbial metabolites (e.g., short-chain fatty acids (SCFA)), regulation of the immune system, and the microbial impact on gut hormones and neurotransmitters. Similarly, intake of fermented foods is positively associated with cognitive health and has been shown to alter the microbiota composition and function and exert an anti-inflammatory effect. However, no studies to date have examined the singular and combined effects of fermented and fibrous foods on the gut microbiota, cognition, and emotion. The present study aims to determine the role of diet on the microbiota-gut-brain axis and mental health.

Using a randomized-controlled, parallel, single-blinded design, participants consuming a habitually low fibre diet (N=200) will undergo an 8-week dietary intervention. Participants will receive one of four diets (n=50 in each group): high fibre (aim 24-35 grams/day), fermented foods (aim 4-6 portions/day), combined diet of fermented foods and high fibre (aim 25-30g/day of fibre and 3-4 servings/day of fermented foods) or control (dietary education according to national Irish guidelines). Cognitive, psychological, and biological measures will be compared at baseline and endpoint. During the intervention period, individuals will provide repeated faecal samples to assess temporal microbial changes.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent.
* Be between 18 and 50 years of age.
* Have a body mass index (BMI) between 18.5-29.9 Kg/m2.
* Be in generally good health as determined by the investigator.

Exclusion Criteria:

* Are less than 18 and greater than 50 years of age.
* Have a BMI below 18.5 or above 29.9 Kg/m2.
* Have a significant acute or chronic coexisting illness [cardiovascular, gastrointestinal (GI) [to include functional GI disorders, inflammatory bowel disease, coeliac disease, lactose intolerance, food allergies], immunological, psychiatric [to include formal or as determined by MINI Psychiatric interview, diagnosis of current major depression, anxiety disorder, bipolar spectrum disorder, schizophrenia, other DSM-IV Axis I disorder], neurodevelopmental disorders, immunological, metabolic disorders [to include type I or II diabetes], or any condition which contraindicates, in the investigators judgement, entry to the study,
* Have a condition or taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk, or confound the interpretation of the study results; all psychoactive medications [to include anxiolytics, antipsychotics, antidepressants, anticonvulsants, centrally acting corticosteroids, and opioid pain relievers), laxatives, enemas, antibiotics, anti-coagulants, over-the counter non-steroidal anti-inflammatories (NSAIDS). Subjects should have a wash-out period of 4 weeks.
* Current prebiotic or probiotic supplement use (a wash-out period of 4 weeks after cessation will allow entry to the study).
* Females who are peri-menopausal, menopausal or post-menopausal.
* Females who are pregnant or planning a pregnancy, or lactating.
* Participants who are not fluent in English.
* Are colour blind.
* Have dyslexia or dyscalculia.
* Are a current habitual daily smoker.
* Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
* Subjects receiving treatment involving experimental drugs. If the subject has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.
* Have a malignant disease or any concomitant end-stage organ disease.
* Have completed a study in our laboratory in the past 4 years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Trait stress/mood: self-report | Change from baseline at 8 weeks
  self-report questionnaires
Trait stress/mood: hypothalamic-pituitary-adrenal axis activity | Change from baseline at 8 weeks
  Cortisol from saliva samples
Responses to acute stress: self-report | Change from baseline at 8 weeks
  Self-report questionnaires
Responses to acute stress: sympathetic-adrenal-medullary pathway activity | Change from baseline at 8 weeks
  Galvanic skin response taken from the skin on the hand
Responses to acute stress: hypothalamic-pituitary-adrenal axis activity | Change from baseline at 8 weeks
  Cortisol from saliva samples

SECONDARY OUTCOMES:
Cognitive performance: working memory | Change from baseline at 8 weeks
  Spatial Working Memory
Cognitive performance: episodic memory | Change from baseline at 8 weeks
  Modified Rey Auditory Verbal Learning Test (ModRey)
Cognitive performance: decision making | Change from baseline at 8 weeks
  Iowa Gambling Task
Cognitive performance: emotional inhibition | Change from baseline at 8 weeks
  Emotional Stroop
Cognitive performance: sustained attention | Change from baseline at 8 weeks
  Rapid Visual Information Processing
Cognitive performance: visual pattern recognition memory | Change from baseline at 8 weeks
  Pattern Recognition Memory
Cognitive performance: cognitive flexibility | Change from baseline at 8 weeks
  Intra-Extra Dimensional Set Shifting
Cognitive performance: social cognition | Change from baseline at 8 weeks
  Emotion Recognition Task
Cognitive performance: affective perceptual bias | Change from baseline at 8 weeks
  Emotional Bias Task
Microbiota composition and function | Change from baseline at 8 weeks
  Shotgun metagenomics of fecal samples
Microbial and host metabolomics | Change from baseline at 8 weeks
  Untargeted metabolomics analysis
Inflammation | Change from baseline at 8 weeks
  Inflammatory markers in lipopolysaccharide stimulated and unstimulated bloods

CONTACTS AND LOCATIONS:
Overall Officials: John Cryan, PhD, Principal Investigator — APC Microbiome Ireland
Locations (1):
- APC Microbiome Ireland, Cork, Ireland